CLINICAL TRIAL: NCT05040035
Title: Influence of Localization of ACT-measurement and Influence of LAA on ACT Among Patients Undergoing Left Atrial Ablation Procedure.
Brief Title: ACT-Measurement at Different Location During Left Atrial Ablation Procedures
Acronym: ACT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Internistisches Klinikum Munchen Sud (Other)
Responsible Party: Sponsor
Other Study IDs: ACT_IKMS_1
Record Dates: First submitted 2021-08-10; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
Keywords: anticoagulation; ablation; atrial fibrillation; ACT
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ACT measurement — Measurement of active clotting time (ACT)

SUMMARY:
Ablation of atrial fibrillation is standard therapy for symptomatic patients or patients with severely reduced systolic left ventricular ejection fraction. Complications of the procedure are ischemic thrombembolic stroke. Therefore periprocedural treatment with heparin is administered to acchieve a therapeutic anticoagulation. The efficacy of anticoagulation is measured by active-clotting time (ACT) which is measured with blood drawn mostly from the V. femoralis.

Despite controlled anticoagulation periprocedural stroke is published with an incidence of up to 2% and asymptomatic cerebral embolization from 2% to 15%.

The ACT-Trial has two aims:

1. Analysis of the influence of the localization of blood drawing on the measured ACT: blood from central venous line, from LA and from LAA.
2. Dependency of the ACT measured in the blood of the LAA with regard to anatomic und functional LAA-measurements.

Patients will be included scheduled for left atrial ablation procedure and will be divided in two groups: atrial fibrillation at time of procedure and sinus rhythm at time of procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 until 80 years with atrial fibrillation scheduled for left atrial ablation procedure (according to 20216 ESC Guidelines for the management of atrial fibrillation" and/or "2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation" 3. signed informed consent. 4. hemoglobin >10 g/dl in Messungen up to 8 weeks before inclusion.

Exclusion criteria:

Incompliance or contraindication of oral anticoagulation prior to ablation procedure.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation scheduled for left atrial ablation procedure
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of mean and median values of ACT measurements from LA und LAA and dependency on anatomic and functional LAA parameters among patients in sinus rhythm. | During ablation procedure
  Active clotting time from left atrium (LA) and left atrial appendage (LAA) measured at the same time.

SECONDARY OUTCOMES:
Target values of ACT measured in central venous line, LA and LAA among patients with sinus rhythm | During ablation procedure
  Active clotting time from left atrium (LA) and left atrial appendage (LAA) measured with regard to target ACT over time during ablation procedure among patients with sinus rhythm.
Target values of ACT measured in central venous line, LA and LAA among patients with atrial fibrillation | During ablation procedure
  Active clotting time from left atrium (LA) and left atrial appendage (LAA) measured with regard to target ACT over time during ablation procedure among patients with atrial fibrillation.
Dynamics of ACT values over time from samples taken from central venous line, LA and LAA among patients with sinus rhythm | During ablation procedure
  Active clotting time from left atrium (LA) and left atrial appendage (LAA) measured with regard to time behaviour during ablation procedure among patients with sinus rhythm.
Dynamics of ACT values over time from samples taken from central venous line, LA and LAA among patients with atrial fibrillation | During ablation procedure
  Active clotting time from left atrium (LA) and left atrial appendage (LAA) measured with regard to time behaviour during ablation procedure among patients with atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Jilek, MD, Principal Investigator — Internistisches Klinikum Munchen Sud; Thorsten Lewalter, Prof, Study Director — Internistisches Klinikum Munchen Sud
Locations (1):
- Internistisches Klinikum München Süd, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No